CLINICAL TRIAL: NCT06594562
Title: Telementored eFAST in Patients Post-Liver Surgery: A Study of Diagnostic Accuracy for Detection of Free Fluid
Brief Title: Free Fluid Detection With Telementored eFAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Brun, Clinical researcher, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 172964
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hemoperitoneum; Ascites; Intra-Abdominal Fluid Collection; Postoperative Complications
Keywords: Teleultrasound; eFAST; Telemedicine; Ultrasound
MeSH Terms: conditions — Hemoperitoneum; Ascites; Postoperative Complications

STUDY DESIGN:
Masking Description: The quality of the teleultrasound images will be assessed by a radiologist who did not participate in the telementoring session, to minimize novelty bias. Additionally, the radiologist conducting the direct examinations will be distinct from the remote expert who provided telementoring, ensuring that they do not rely on prior knowledge from the remote sessions. While no formal masking will be implemented, these measures are taken to reduce potential bias in the assessment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telementored eFAST (Experimental): Ultrasound examination guided in real-time by a remote expert for detecting free fluid, compared to standard ultrasound performed by on-site radiologist.
  Interventions: Diagnostic Test: Telementored eFAST

INTERVENTIONS:
Diagnostic Test: Telementored eFAST — Ultrasound examination guided in real-time by a remote expert for detecting free fluid.

SUMMARY:
This feasibility study will evaluate the accuracy of telementored eFAST (Extended Focused Assessment with Sonography in Trauma) in detecting abdominal free fluid in patients who have recently undergone liver surgery. The primary goal is to determine how well the remote-guided ultrasound can identify fluid accumulation compared to conventional ultrasound performed by a radiologist. Participants in this study will be examined with ultrasound, supported in real-time by a remote expert, to assess its accuracy and other relevant performance metrics.

DETAILED DESCRIPTION:
The study is designed as a prospective diagnostic trial and involves 40 patients at Oslo University Hospital.

Participants will receive an ultrasound examination shortly after surgery, where a nurse is guided in real-time by a remote expert via teleultrasound. The primary objective is to assess the agreement between the telementored eFAST examination and a conventional ultrasound performed by an on-site radiologist. In addition to diagnostic accuracy, the study will evaluate various performance metrics, including the duration of the telementored versus conventional examinations, network reliability, and cognitive workload using the NASA Task Load Index.

The study will also explore the learning curve associated with telementored eFAST by monitoring the improvement in examination efficiency over time. These metrics will help determine the feasibility of using telementored ultrasound as a reliable diagnostic tool in postoperative care, potentially reducing the need for more resource-intensive imaging modalities and improving patient outcomes through timely decision-making.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone laparoscopic liver surgery at the Oslo university hospital and are within 72 post-surgery

Exclusion Criteria:

Allergy to ultrasound gel. Patients colonized with ESBL, MRSA and VRE will be excluded due to infection control. Significant postoperative pain that can exacerbated by probe pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Concordance rate | Assessed immediately after each ultrasound examination (telementored and conventional) for each participant
  Comparison of telementored eFAST vs. CT and expert examination with percentage agreement
Exam duration | Within 72 hours of surgery for each participant
  Time measurement from probe contact to mutual agreement between expert and examiner that exam is finished in minutes:seconds
Image quality | Assessed retrospectively at the end of data collection, expected to be within 6 months after the final recorded examination
  An independent radiologist will assess the image quality using a 1-5 Likert scale based on a feedback questionnaire adapted from Mazur et al

SECONDARY OUTCOMES:
Mental effort | Immediately after each telementored eFAST examination
  Cognitive workload during eFAST, measured by NASA Task Load Index on a numerical score (1-9)
User experience | Immediately after each telementored eFAST examination
  Feedback questionnaire adapted from McBeth et al.
Learning curve (Mental effort) | Data will be evaluated cumulatively at the end of the study, through study completion, estimated to be up to 6 months after the final participant's examination
  Asess improvement in eFAST exam efficiency by comparing mental effort over multiple examinations
Learning curve (efficiency) | Assessed cumulatively through study completion, estimated up to 6 months after final participant examination
  Evaluate whether telementored examiners show changes in eFAST examination duration over time. The duration of each examination will be compared to previous ones for the same examiner to identify trends in efficiency across multiple sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Brun, Professor, Study Director — Oslo University Hospital
Locations (1):
- Oslo university hospital, Rikshospitalet, Oslo, Oslo County, Norway